CLINICAL TRIAL: NCT04496323
Title: Physical Activity and Energy Expenditure in Golf
Brief Title: Energy Expenditure in Golf
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: EE_Golf
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Physical activity; Golf; Exercise; Energy consumption; METs
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LOW: Golf Skill level high, handicap below 11.5
  Interventions: Other: EE Golf
- HIGH: Golf Skill level low, handicap 18.5 - 26.4
  Interventions: Other: EE Golf

INTERVENTIONS:
Other: EE Golf — Exercise in Golf and Playing 9 holes

SUMMARY:
Structured exercise and physical activity are well known to not only improve physical fitness, but also alter various health parameters in a positive fashion. To yield health benefits, exercises need to meet certain characteristics e. g. specific levels of intensity or duration.To evaluate intensity levels and therefor possible improvements in physical conditioning in golf the investigators conducted this study with two groups of each 10 subjects. The groups differed in age and skill level (handicap, hcp). Each group went through a exercise session on the driving range (DR) and a 9-hole compeition round of golf. The investigators assessed spirometrical data (breath-by-breath) to evaluate energy expenditure (EE) and intensity levels of physical activity according to the ACSM guidelines.

ELIGIBILITY:
Inclusion Criteria:

* male
* age 18 to 45 y
* Body-Mass-Index: under 30 kg/m2
* Handicapclasses 1,2 und 4
* healthy

Exclusion Criteria:

* contraindication (orthopaedic, cardiologic, etc.) to participating in physical exhausting force and endurance testing and playing golf
* acute or chronical inflammation
* intake of drugs and medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Members of German golf clubs with an active playing status.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Metabolic Äquivalent of Task (MET) | 90 minutes
  1 MET = 3.5 mL of oxygen per kilogram bodyweight per minute

SECONDARY OUTCOMES:
Percent Heart Rate | 90 minutes
  Heartrate in in relation to maximum heartrate
Percent VO2 | 90 minutes
  oxygen uptake in relation maximum oxygen uptake (VO2peak)
Duration of Intensity levels in METs | 90 minutes
  Relative time spent in intensity levels

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Tegtbur, Prof., Study Director — Hannover Medical School

IPD SHARING:
Plan to Share IPD: Undecided